CLINICAL TRIAL: NCT06660706
Title: The Effects of Exercise Intervention on Skeletal Muscle and Other Organs in Aged Population and the Discovery of Associated Circulating Biomarkers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Principal Investigator, Li-Ning Peng, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NYCU112162AF
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Age-related Functional Decline
Keywords: aging; muscle health; body composition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multidomain intervention group (Experimental): The multidomain intervention program is designed as structural training sessions of 2-hour training sessions two times per week.
  Interventions: Behavioral: Multi-domain intervention
- Usual care group (No Intervention): Provide conventional health educations in every three-month interval

INTERVENTIONS:
Behavioral: Multi-domain intervention — Each session comprises of 45 minutes physical fitness activities targeting on muscle strength, balance, and flexibility; 1-hour cognitive training primarily on reasoning and memory exercises; and 15-minute for nutritional advices based on national diet guidelines for older adults
  Arms: Multidomain intervention group

SUMMARY:
This project aims to investigate the intricate interplay between skeletal muscle and adipose tissue during the aging process by integrating human studies. Utilizing interventional research and randomized trials combined with examining blood samples from elderly individuals engaged in exercise, we aim to investigate the effects of exercise on muscle health and explore the underlying mechanisms of muscle aging and related biomarkers. Interdisciplinary research allowed us to investigate the systemic impact of exercise on muscles. This approach allowed us to gain a better understanding of the interconnectedness of skeletal muscle and adipose tissue in the aging process and devise efficient strategies to reverse age-related changes. These findings hold promise for promoting a future society where long and healthy life is achievable for all.

DETAILED DESCRIPTION:
This study is a randomized controlled trial of 6-month multidomain intervention program among community-living older adults with early physical impairments.

Inclusion criteria are: (1) community-dwelling adults aged ≥ 65 years, (2) slow gait speed (<1 m/s in 6-meter walk test) or weakness (dominant handgrip strength <28 kg in men, <18 kg in women); subjects with the following conditions will be excluded: (1) established diagnosis of dementia, Parkinsonism or other neurodegenerative disease (2) disable status: mobilitylimiting conditions, (3) active, acute diseases receiving treatment, such as cancer, heart failure, COPD and so on, (4) estimated life expectancy <12 months, (5) current nursing home residents.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 65 years
* slow gait speed (<1 m/s in 6-meter walk test) or weakness (dominant handgrip strength <28 kg in men, <18 kg in women)

Exclusion Criteria:

* established diagnosis of dementia, Parkinsonism or other mobility-limiting, disable conditions
* active, acute diseases receiving treatment, such as cancer, heart failure, COPD and so on
* estimated life expectancy <12 months
* current nursing home residents

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Physical performance | baseline, 6 month
  Change in hand-grip strength (kg), or six-meter walking speed (m/s), or 5 times sit to stand test from baseline to 6 months in all participants

SECONDARY OUTCOMES:
Change in DHEA-S | baseline, 6 month
  Change in DHEA-S concentration from baseline to 6 months in all participants
Change in IGF-1 | baseline, 6 month
  Change in IGF-1 concentration from baseline to 6 months in all participants
Change in hs-CRP | baseline, 6 month
  Change in hs-CRP concentration from baseline to 6 months in all participants
Change in Myostatin | baseline, 6 month
  Change in Myostatin concentration from baseline to 6 months in all participants
Change in Activing A | baseline, 6 month
  Change in Activing A concentration from baseline to 6 months in all participants
Change in Follistatin | baseline, 6 month
  Change in Follistatin concentration from baseline to 6 months in all participants
Change in Relative appendicular skeletal muscle index (RASM) | baseline, 6 month
  Change in RASM from baseline to 6 months in all participants
Change in body fat % | baseline, 6 month
  Change in body fat % from baseline to 6 months in all participants
Change in Cognitive performance | baseline, 6 month
  Change in Montreal Cognitive Assessment (MoCA), or Mini-mental state examination (MMSE) from baseline to 6months in all participants
Change from lipoproflie | baseline, 6 month
  Change in Total Cholesterol, Triglyceride, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol from baseline to 6months in all participants

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ning Peng, M.D., PhD, Principal Investigator — Center for Healthy Longevity and Aging Sciences, National Yang Ming Chiao Tung University
Locations (1):
- Center for Healthy Longevity and Aging Sciences, National Yang Ming Chiao Tung University, Taipei, Taiwan